CLINICAL TRIAL: NCT07064577
Title: Novel ROS-scavenging Nanoenzymes for the Treatment of Radiation Dermatitis in Patients With Head and Neck Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024-134-1
Record Dates: First submitted 2025-07-11; First posted 2025-07-14 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Radiation Dermatitis
MeSH Terms: conditions — Radiodermatitis | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ROS-scavenging Nanoenzymes (Experimental)
  Interventions: Drug: ROS-scavenging Nanoenzymes
- Standard of care (Active Comparator)
  Interventions: Behavioral: Standard of care

INTERVENTIONS:
Drug: ROS-scavenging Nanoenzymes — ROS-scavenging nanoenzymes are applied to the treatment area, once daily during radiotherapy.
  Arms: ROS-scavenging Nanoenzymes
Behavioral: Standard of care — Standard of care
  Arms: Standard of care

SUMMARY:
There is no standard treatment for radiation dermatitis. In this study, the investigators have designed novel ROS-scavenging nanoenzymes and aim to evaluate their effectiveness in preventing radiation dermatitis in patients with head and neck cancer.

DETAILED DESCRIPTION:
Radiotherapy often leads to various complications, with radiation dermatitis being the most common side effect observed in the majority of tumor patients undergoing treatment. This condition not only affects a patient's appearance but, in severe cases, may even require the interruption of treatment.

Currently, there is no standard treatment for radiation dermatitis. In this study, the investigators have designed novel ROS-scavenging nanoenzymes, offering a potential new approach for preventing and treating radiation dermatitis.

This clinical trial aims to evaluate the effectiveness of these novel ROS-scavenging nanoenzymes in preventing radiation dermatitis in patients with head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a pathological diagnosis of non-metastatic head and neck malignant tumors;
2. Patients deemed suitable for high-dose radiotherapy, either as a primary treatment or as postoperative treatment following surgical resection.

Exclusion Criteria:

1. Eastern Cooperative Oncology Group performance status of >2;
2. Pre-existing skin rash, ulceration or open wound in the treatment area;
3. Inflammatory or connective tissue disorder of the skin;
4. History of head and neck radiotherapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
The incidence of grade 2 or higher radiation dermatitis | From the start of radiotherapy to 2 weeks after completion of radiotherapy.
  Patients are assessed weekly for radiation dermatitis by an experienced radiation oncology nurse according to the Radiation Therapy Oncology Group (RTOG) criteria.

SECONDARY OUTCOMES:
The maximum skin toxicity | From the start of radiotherapy to 2 weeks after completion of radiotherapy.
  The maximum grade of RTOG skin toxicity between 0 and 4.

CONTACTS AND LOCATIONS:
Overall Officials: Xingchen Peng, Prof., Principal Investigator — Sichuan University West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No